CLINICAL TRIAL: NCT02790736
Title: Brief Intervention to Reduce Fear of Public Speaking
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 restrictions
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Franklin Schneier, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 7293 (SAD); NCT02924610 (obsolete NCT alias)
Record Dates: First submitted 2016-05-26; First posted 2016-06-06 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: Social Anxiety Disorder
Keywords: propranolol; public speaking anxiety
MeSH Terms: conditions — Phobia, Social | interventions — Propranolol; propranolol CR

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propranolol (Experimental): Propranolol 40 mg capsule, given once after fear activation procedure
  Interventions: Drug: propranolol
- placebo capsule (Placebo Comparator): Placebo capsule, given once after fear activation procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: propranolol — active treatment
  Other Names: Innopran XL
  Arms: Propranolol
Drug: Placebo — inactive pill
  Other Names: Placebo Oral Tablet
  Arms: placebo capsule

SUMMARY:
The study will test the efficacy of propranolol or placebo, administered after retrieval of a previously acquired public speaking fear, in reducing fear and avoidance of public speaking.

DETAILED DESCRIPTION:
Twenty subjects with Performance-Only type of Social Anxiety Disorder will be enrolled in the study. Participants will complete baseline assessments of fear and avoidance of public speaking. Participants will be randomly assigned to a single dose of propranolol 40mg or placebo, administered immediately after a fear activation procedure. Primary outcome assessment will be self-reported fear of public speaking and avoidance behavior in a behavioral avoidance task 2 weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age at the time of consent
* Principal Diagnosis of Social Anxiety Disorder, Performance only type
* Has clinically significant fear of public speaking
* Physically healthy
* If female, non-pregnant and not nursing
* Off all psychotropic drug for at least 4 weeks
* A level of understanding sufficient to provide written informed consent to all required study tests and procedures.

Exclusion Criteria:

* History of other serious psychiatric disorder
* Current Major Depressive Disorder
* Presence of developmental disorder or intellectual disability
* SAD patients with SAD not of the performance only type
* Women who are pregnant or nursing
* Current use of psychiatric medication
* Current substance use disorder
* Persons planning to start another treatment during the study period.
* Any significant medical condition that might increase the risk or participation (e.g., seizure disorder, respiratory disorders [e.g., bronchial asthma], cardiovascular disease [e.g., congestive heart failure, heart arrhythmias, sinus bradycardia and greater than first degree block ], low blood pressure [ < 90/60], diabetes, liver or kidney disorders)
* Use of medications that might negatively interact with propranolol (e.g., ACE inhibitors; catecholamine depleting drugs, such as reserpine; calcium channel blockers; digitalis glycosides; haloperidol; chlorpromazine; aluminum hydroxide gel; phenytoin; phenobarbitone; rifampin; antipyrine; lidocaine; cimetidine; theophylline)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Study Director — NYSPI
Locations (1):
- New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Propranolol | Placebo Capsule
Started | 5 | 1
Completed | 5 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propranolol | Placebo Capsule | Total
Number analyzed (Participants) | 5 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Personal Report of Confidence as a Speaker
Description: total score on this self report measure of fear of public speaking. Scored from 0-30, with higher scores indicating better outcome
Time Frame: 2 weeks
Population: persons with fear of public speaking
Measure: Mean (Full Range); unit: change score on a scale
Arm/Group | Propranolol | Placebo Capsule
Number analyzed (Participants) | 5 | 1
change score on a scale | 6.6 [1 to 13] | 6 [6 to 6]

2. Secondary Outcome: Behavioral Avoidance Task
Description: Up to 5 sequential public speaking challenges, specifically designed for each step to be of increasing difficulty for the individual. Each step is considered completed if subject agrees to try speaking, and speaks for 1 minute. Score is total number of completed steps (0-5) on this 5-step task, with 5 being best
Time Frame: 2 weeks
Measure: Mean (Full Range); unit: steps
Arm/Group | Propranolol | Placebo Capsule
Number analyzed (Participants) | 5 | 1
steps | 4.2 [4 to 5] | 4 [4 to 4]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Propranolol | Placebo Capsule
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/1
Other Adverse Events (participants affected / at risk) | 0/5 | 0/1

LIMITATIONS AND CAVEATS:
Early termination of this pilot study leading to small numbers of subjects evaluated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT02790736/Prot_SAP_ICF_000.pdf